CLINICAL TRIAL: NCT03809520
Title: An Imaging Framework for Clinically Testing New Treatments to Prevent Post-traumatic OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: J L Marsh (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor-Investigator, J L Marsh, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201612747
Record Dates: First submitted 2018-12-20; First posted 2019-01-18 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Orthopedic Disorder; Trauma; Ankle Fractures; Post-traumatic Osteoarthritis
MeSH Terms: conditions — Musculoskeletal Diseases; Wounds and Injuries; Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental: pedCAT (Experimental): Subjects in this group will undergo weight-bearing CT (pedCAT) imaging at 6 months, 12 months, and 18 months post-ankle injury.
  Interventions: Radiation: pedCAT

INTERVENTIONS:
Radiation: pedCAT — Weight-bearing CT scan (pedCAT) of ankles to measure 3D joint space width following ankle fracture.

SUMMARY:
The immediate goal of the proposed research is to test the value of a new low-cost, low-dose standing CT system for efficient early detection of both joint degeneration and elevated contact stress. The standing CT scanner holds promise for detecting arthritic changes earlier than other imaging modalities because of the combination of its 3D nature and ability to image joints in a weight-bearing pose. A secondary goal of the proposed research is to enable predictive models for osteoarthritis risk based on measures of post treatment contact stress, both to inform treatment and so that new interventions can be tested in a manner incorporating risk stratification.

DETAILED DESCRIPTION:
Individuals who present with an intra-articular of the tibial plafond will be consented to participate in this study. We will obtain pedCAT scans at 6, 12, and 18 months post-injury, as well as several questionnaires that will be administered during the clinical visits. We will also review the subjects' electronic medical record for data related to the injury, including the timing and mechanism of injury, time from injury to surgery, length of hospital stay, any complications and/or subsequent ankle surgeries, as well as any clinic notes, imaging, and/or outcomes scores related to the calcaneus fracture.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 to 70 years old Sustained an intra-articular fracture of the tibial plafond Indicated for operative treatment Present for treatment within 4 weeks of injury

Exclusion Criteria:

* Women who are pregnant or planning on becoming pregnant Individuals younger than 18 and older than 70

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the ankle joint space width | 18 months
  Tracking longitudinal changes in the 3D joint space width as seen in pedCAT imaging compared to baseline pedCAT imaging

SECONDARY OUTCOMES:
Change in ankle pain | 18 months
  Subjective measure of foot and ankle pain gathered by patient reported outcomes questionnaires
Change in ankle function | 18 months
  Subjective measure of foot and ankle function gathered by patient reported outcomes questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: J L Marsh, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No